CLINICAL TRIAL: NCT06167031
Title: The Effectiveness of Chatbot Facilitated Education on Child and Adolescent Abuse for Nurses
Brief Title: Chatbot Facilitated Education on Child and Adolescent Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Li-Cheng Kao, RN, MSN, Co-Project Investigator, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB112-148-B
Record Dates: First submitted 2023-10-05; First posted 2023-12-12 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Child Abuse
Keywords: child and adolescent abuse and neglect (CAAN); chatbots; attitude toward reporting; intention to report

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot-facilitated education Group (Experimental): The participants will receive a lecture on the CAN course with assistance from a chatbot. The instructor will pose questions to the participants, who will respond using the chatbot.
  Interventions: Other: chatbot facilitated teaching
- Lecture-based teaching Group (Active Comparator): The participants will only receive a lecture on the CAN course.
  Interventions: Other: lecture-based teaching

INTERVENTIONS:
Other: chatbot facilitated teaching — The experimental group will use "chatbot" to facilitate teaching.
  Arms: Chatbot-facilitated education Group
Other: lecture-based teaching — The control group only receives lecture-based teaching.
  Arms: Lecture-based teaching Group

SUMMARY:
The study aims to evaluate the effectiveness of chatbot-facilitated education (CFE) in assisting nursing personnel to prevent child and adolescent abuse and neglect (CAN). The main questions it aims to answer are:

1. Does applying CFE enhance nurses' intention to report CAN?
2. Does applying CFE improve nurses' attitudes toward reporting CAN?
3. Does applying CFE increase nurses' knowledge of CAN?

Researchers will compare CFE to lecture-based teaching to verify if CFE can improve the nurses' competency of CAN.

Participants will:

1. Attend a CAN course for about 1.5 hours. The experimental group will use CFE, and the control group will only receive lecture-based teaching.
2. Have the CAN course, comprised of two main subjects: "CAN" and "Nurses' Roles and Functions in CAN".
3. Receive the learning effect assessment at three different time points: before the course, one week after, and four weeks after.

DETAILED DESCRIPTION:
Based on the rigor of the study and the anticipated benefits to the participants, we will:

1. Commence participant enrollment only after the protocol has been reviewed and approved by the Research Ethics Committee of Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation.
2. Conduct a minimum of four courses until the participant group reaches full capacity.
3. Ensure that participants are not informed about the specific interventions of the course at the time of their enrollment.

ELIGIBILITY:
Inclusion Criteria:

Nurses who

1. work in Hualien Tzu Chi Hospital
2. finish the probationary period, directly do the practical care
3. want to participate and sign the consent

Exclusion Criteria:

The nurses will be excluded if they are in an administrative position or withdraw the protocol for any reason.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Lin Hsieh, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, Hualien County, Taiwan

IPD SHARING:
Plan to Share IPD: No
Our study won't share the IPD with others. It has been written on the participants' consent.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled the participants for a year from July 2023 at a tertiary hospital in eastern Taiwan.
Pre-assignment Details: Course promotion commenced in July 2023. The first participant was not enrolled until the inaugural course launched on January 10, 2024. During the six-month preparatory period, we engaged in iterative planning, instructional design, and repeated testing of both the course delivery system and the integrated chatbot functionality.
Groups:
- Chatbot-facilitated Education Group: Chatbot facilitated teaching: The experimental group will use "chatbot" to facilitate lecture-based teaching.
Period: Overall Study
Arm/Group | Chatbot-facilitated Education Group | Lecture-based Teaching Group
Started | 49 | 49
Completed | 44 (The participants who have finished two post-tests are defined as completed.) | 48 (The participants who have finished two post-tests are defined as completed.)
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Population: Five participants in the experimental group and one in the control group didn't finish either post-test one or two. So they couldn't be included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chatbot-facilitated Education Group | Lecture-based Teaching Group | Total
Number analyzed (Participants) | 44 | 48 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.4) | 29.2 (7.0) | 28.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 4 | 9 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Job tenure [Mean (Standard Deviation); unit: years] | 5.2 (5.1) | 6.0 (6.2) | 5.6 (5.7)
Units [Count of Participants; unit: Participants]
  Emergency depaertment | 15 | 17 | 32
  Pediatric | 10 | 2 | 12
  Medical Surgical Unit | 14 | 24 | 38
  Adult intensive care units | 5 | 5 | 10
Level of nursing [Count of Participants; unit: Participants] — According to the Taiwan Nurses Association, clinical nurses are classified into five levels:
  N - Less than 1 year of experience; N1 - At least 1 year of experience and able to provide basic patient care; N2 - 2 years of experience and competent in caring for critically ill patients; N3 - 3 years of experience with the ability to deliver holistic critical care, teach, and support quality improvement; N4 - 4 years of experience, responsible for advanced critical care, teaching, administration, and unit-based quality initiatives.
  Participants
    N | 9 | 18 | 27
    N1 | 8 | 5 | 13
    N2 | 18 | 16 | 34
    N3 | 9 | 9 | 18
    N4 | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Associate Degree | 3 | 7 | 10
  Bachelor's Degree | 41 | 41 | 82
  Master's Degree | 0 | 0 | 0
  Doctorate (Ph.D.) | 0 | 0 | 0
The experience of dealing with child and adolescent abuse and neglect [Count of Participants; unit: Participants]
  Yes | 26 | 22 | 48
  No | 18 | 26 | 44
The experience of receiving training in child and adolescent abuse and neglect [Count of Participants; unit: Participants]
  Yes | 14 | 17 | 31
  No | 30 | 31 | 61
The experience of receiving education by using a chatbot [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 43 | 48 | 91
The motives for participating [Count of Participants; unit: Participants]
  Interest | 19 | 20 | 39
  Required competency in the workplace | 11 | 14 | 25
  Assignment of workplace | 1 | 1 | 2
  Requirement of nursing credits | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Intention to Report Child and Adolescent Abuse and Neglect
Description: This subscale is part of the Child and Adolescent Abuse and Neglect (CAN) Competency Assessment. It comprises eight simulated child abuse scenarios, with participants rating their intention to report each case on an 11-point scale ranging from 0 (no intention to report) to 10 (definite intention to report). The total possible score is 80, with higher scores indicating a stronger and more consistent intention to report suspected CAN cases.
Time Frame: Pre-test (before the course), Post-test 1 (one week after), Post-test 2(four weeks after).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chatbot-facilitated Education Group | Lecture-based Teaching Group
Number analyzed (Participants) | 44 | 48
score on a scale
  Pre-test | 60.77 (10.11) | 61.56 (10.41)
  Post-test 1 | 71.07 (6.51) | 68.29 (8.91)
  Post-test 2 | 69.34 (11.77) | 68.73 (8.81)

2. Primary Outcome: Attitude Toward Reporting Child and Adolescent Abuse and Neglect
Description: This subscale is part of the Child and Adolescent Abuse and Neglect (CAN) Competency Assessment and consists of three sections: five items on attitudes toward child discipline, six items on perceptions of abusive parents, and seven items on professional responsibility in reporting child abuse, totaling 18 items. Participants rate each item on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree). The maximum possible score is 108. Higher scores reflect more negative attitudes toward physical discipline, lower tolerance for abusive behavior by parents, and stronger endorsement of professional responsibility in reporting suspected child abuse.
Time Frame: Pre-test (before the course), Post-test 1 (one week after), Post-test 2(four weeks after).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chatbot-facilitated Education Group | Lecture-based Teaching Group
Number analyzed (Participants) | 44 | 48
score on a scale
  Pre-test | 83.52 (8.72) | 82.40 (8.69)
  Post-test 1 | 84.70 (9.50) | 82.19 (8.53)
  Post-test 2 | 85.14 (9.08) | 80.73 (11.0)

3. Primary Outcome: Knowledge About Child and Adolescent Abuse and Neglect
Description: This subscale is part of the Child and Adolescent Abuse and Neglect (CAN) Competency Assessment and includes 13 true-false items. Participants are instructed to respond with "true," "false," or "don't know" for each statement. Correct responses receive one point, while incorrect or "don't know" responses receive zero. The total possible score is 13, with higher scores indicating greater knowledge of CAN and its relevant legal framework.
Time Frame: Pre-test (before the course), Post-test 1 (one week after), Post-test 2(four weeks after).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chatbot-facilitated Education Group | Lecture-based Teaching Group
Number analyzed (Participants) | 44 | 48
score on a scale
  Pre-test | 7.95 (2.12) | 8.75 (1.79)
  Post-test 1 | 9.66 (1.70) | 9.52 (1.86)
  Post-test 2 | 9.32 (1.89) | 9.29 (2.06)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants were instructed to report any adverse events during the study. However, the intervention involved only a didactic course and access to a chatbot delivered via participants' personal mobile phones. No adverse events were reported throughout the study period.
Arm/Group | Chatbot-facilitated Education Group | Lecture-based Teaching Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT06167031/Prot_SAP_000.pdf